CLINICAL TRIAL: NCT01275651
Title: Androgen Receptor (AR) Activity in Castration-Resistant Prostate Cancer (CRPC) and Response to Ketoconazole
Brief Title: Biomarkers in Bone Marrow and Blood Samples From Patients With Prostate Cancer Treated With Ketoconazole
Status: Withdrawn | Type: Observational
Why Stopped: Trial closure for NCI NCTN Transition
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-151004; CDR0000688286 (Registry Identifier: NCI Physician Data Query); NCI-2011-02835 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue, bone marrow, and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (AR activity in CRPC): Previously collected bone marrow tissue and blood samples are analyzed for AR activity, AR splice variations, expression of androgen transport/synthesis/metabolism genes, AKR1C3 protein levels, and testosterone and dihydrotestosterone levels via RT-PCR, SNP microarrays, IHC, gene expression analysis, and mass spectrometry methods.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies biomarkers in bone marrow and blood samples from patients with prostate cancer treated with ketoconazole. Studying samples of bone marrow and blood from patients with prostate cancer in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether pre-treatment androgen receptor (AR) activity correlates with progression-free survival (PFS) of men with castration-resistant prostate cancer (CRPC) treated with ketoconazole.

SECONDARY OBJECTIVES:

I. To determine if expression of androgen transport/synthesis/metabolism genes (including cytochrome P450, family 17, subfamily A, polypeptide 1 [CYP17A1], aldo-keto reductase family 1 [AKR1]C3, hydroxy-delta-5-steroid dehydrogenase, 3 beta- and steroid delta-isomerase 2 [HSD3B2], hydroxysteroid [17-beta] dehydrogenase [HSD17B]3, HSD17B6, AKR1C2, AKR1C1, UGTB15, UGTB17, steroid-5-alpha-reductase, alpha polypeptide 1 [3-oxo-5 alpha-steroid delta 4-dehydrogenase alpha] [SRD5A]1, SRD5A2, SRD5A3, and solute carrier organic anion transporter family, member 2B1 [SLCO2B1]) correlate with detected AR activity, time to progression (progression free survival [PFS]) following treatment with ketoconazole, and overall survival.

II. To determine if semi-quantitative immunohistochemical analysis of AR and AKR1C3 protein levels correlate with PFS following treatment with ketoconazole.

III. To determine if specific AR splice variations correlate with PFS in response to ketoconazole.

IV. To determine if detected activity of signaling pathways that interact with AR pathway activity (e.g., phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha [PI3K] and downstream effectors, SRC proto-oncogene, non-receptor tyrosine kinase [SRC], others) correlate with detected AR activity, PFS, and OS.

V. To determine if AR gene amplification correlates with detected AR activity and PFS on ketoconazole.

VI. To determine if levels of testosterone and dihydrotestosterone (DHT) from tumor tissue correlate with AR activity and PFS on ketoconazole.

VII. To determine the presence of specific prostate cancer-associated gene translocations in each sample of CRPC.

VIII. To provide an unbiased data set of gene expression in CRPC that will markedly expand the currently available public domain data.

IX. To provide a library of amplified ribonucleic acid (RNA) and complementary (c)DNA for further analysis by other investigators.

OUTLINE:

Previously collected bone marrow, tissue, and blood samples are analyzed for AR activity, AR splice variations, expression of androgen transport/synthesis/metabolism genes, AKR1C3 protein levels, and testosterone and dihydrotestosterone levels via reverse transcription (RT)-polymerase chain reaction (PCR), single nucleotide polymorphisms (SNP) microarrays, immunohistochemistry (IHC), gene expression analysis, and mass spectrometry methods.

ELIGIBILITY:
Inclusioin Criteria:

* Patients must have been registered to CALGB 9583 and CALGB 9663
* Adequate tissue specimen available for analysis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with prostate cancer registered to Cancer and Leukemia Group B (CALGB) 9583 and CALGB 9663
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Baseline

SECONDARY OUTCOMES:
Equal to or greater than 30% decline in PSA | Baseline
Overall survival | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Study Chair — Dana-Farber Cancer Institute
Locations (1):
- Alliance for Clinical Trials in Oncology, Boston, Massachusetts, United States